CLINICAL TRIAL: NCT03165864
Title: A Double-Blind, Placebo-Controlled, Dose-Escalation, Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Doses of ISIS 702843 Administered Subcutaneously to Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ISIS 702843 Administered Subcutaneously to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 702843-CS1
Record Dates: First submitted 2017-05-18; First posted 2017-05-24 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Thalassemia
Keywords: Thalassaemia, IONIS TMPRSS6-Lrx
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IONIS TMPRSS6-Lrx (Experimental): Ascending single and multiple doses of IONIS TMPRSS6-Lrx administered subcutaneously
  Interventions: Drug: IONIS TMPRSS6-Lrx
- Placebo (Placebo Comparator): Saline .9%
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: IONIS TMPRSS6-Lrx — Ascending single and multiple doses of IONIS TMPRSS6-Lrx administered subcutaneously
  Arms: IONIS TMPRSS6-Lrx
Other: Placebo — Saline .9%
  Arms: Placebo

SUMMARY:
The purpose is to assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IONIS TMPRSS6-Lrx Administered Subcutaneously for up to 44 Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Must have given written informed consent and be able to comply with all study requirements
* Healthy males or females aged 18-65 inclusive at the time of Informed Consent
* Females must be non-pregnant and non-lactating, and either surgically sterile or post- menopausal
* Males must be surgically sterile, abstinent or using an acceptable contraceptive method
* BMI < 32 kg/m2

Exclusion Criteria:

* Clinically significant abnormalities in medical history or physical examination
* Clinically significant lab abnormalities that would render a subject unsuitable for inclusion
* Known history or positive test for HIV, HCV, or HBV
* Treatment with another Study Drug, biological agent, or device within one-month of Screening or 5 half-lives of investigational agent, whichever is longer
* Smoking > 10 cigarettes per day
* Regular excessive use of alcohol within 6 months of screening
* Current use of concomitant medications other than occasional acetaminophen (paracetamol) or ibuprofen unless approved by Sponsor Medical Monitor
* Considered unsuitable for inclusion by the Investigator or Sponsor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events that are related to treatment with IONIS TMPRSS6-Lrx | Up to 148 Days
  The safety and tolerability of single and multiple doses of IONIS TMPRSS6-Lrx will be assessed by determining the incidence, severity, and dose relationship of adverse events that are related to treatment with IONIS TMPRSS6-Lrx

SECONDARY OUTCOMES:
Pharmacokinetics after single and multiple doses of IONIS TMPRSS6-Lrx (maximum observed drug concentration or Cmax) | Up to 148 Days
  The plasma pharmacokinetics (maximum observed drug concentration or Cmax) of Ionis TMPRSS6-Lrx will be assessed following single and multiple dose SC administration
Pharmacokinetics after single and multiple doses of IONIS TMPRSS6-Lrx (time taken to reach maximal concentration or Tmax) | Up to 148 Days
  The plasma pharmacokinetics (time taken to reach maximal concentration or Tmax) of Ionis TMPRSS6-Lrx will be assessed following single and multiple dose SC administration
Pharmacokinetics after single and multiple doses of IONIS TMPRSS6-Lrx (Plasma terminal elimination half-life (t1/2λz) | Up to 148 Days
  The plasma pharmacokinetics (Plasma terminal elimination half-life (t1/2λz) of Ionis TMPRSS6-Lrx will be assessed following single and multiple dose SC administration
Pharmacokinetics after single and multiple doses of IONIS TMPRSS6-Lrx (Partial areas under the plasma concentration-time curve from zero time (predose) to selected times (t) after the subcutaneous administration (AUCt) | Up to 148 Days
  The plasma pharmacokinetics (Partial areas under the plasma concentration-time curve from zero time (predose) to selected times (t) after the subcutaneous administration (AUCt) of Ionis TMPRSS6-Lrx will be assessed following single and multiple dose SC administration
Pharmacokinetics after single and multiple doses of IONIS TMPRSS6-Lrx (Percentage of the administered dose excreted in urine (% Dose Excreted) | Up to 148 Days
  The plasma pharmacokinetics (Percentage of the administered dose excreted in urine (% Dose Excreted) of Ionis TMPRSS6-Lrx will be assessed following single and multiple dose SC administration

OTHER OUTCOMES:
Pharmacodynamics after single and multiple doses of IONIS TMPRSS6-Lrx (Changes in transferrin saturation) | Up to 148 Days
  Effects of IONIS TMPRSS6-Lrx on changes (absolute and percent) in transferrin saturation compared to baseline
Pharmacodynamics after single and multiple doses of IONIS TMPRSS6-Lrx (Changes in serum iron) | Up to 148 Days
  Effects of IONIS TMPRSS6-Lrx on changes (absolute and percent) in serum iron compared to baseline
Pharmacodynamics after single and multiple doses of IONIS TMPRSS6-Lrx (Changes in hepcidin levels) | Up to 148 Days
  Effects of IONIS TMPRSS6-Lrx on changes (absolute and percent) in hepcidin levels compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Ganz T, Nemeth E, Rivella S, Goldberg P, Dibble AR, McCaleb ML, Guo S, Monia BP, Barrett TD. TMPRSS6 as a Therapeutic Target for Disorders of Erythropoiesis and Iron Homeostasis. Adv Ther. 2023 Apr;40(4):1317-1333. doi: 10.1007/s12325-022-02421-w. Epub 2023 Jan 23. PMID 36690839